CLINICAL TRIAL: NCT06024681
Title: Investigating the Impact of Faecal Microbiota Transplant on the Clinical Phenome of Patients With Non-alcoholic Fatty Liver Disease and Fibrosis
Brief Title: Impact of FMT on the Phenome in Patients With NAFLD and Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ICL_21SM6787; 296522 (Other: IRAS); 21/LO/0454 (Other: REC)
Record Dates: First submitted 2023-08-23; First posted 2023-09-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Fecal Microbiota Transplantation
Keywords: NAFLD; Gut microbiome; Metabolomics
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Human participants with NAFLD and fibrosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NAFLD patients (Experimental): Patients receiving capsulised FMT
  Interventions: Other: Faecal microbiota transplant

INTERVENTIONS:
Other: Faecal microbiota transplant — Capsulised faecal microbiota transplant prepared from rationally selected donor, based upon donor metabolomic charateristics

SUMMARY:
The goal of this pilot experimental medicine interventional study is to explore the degree of transferability of the gut microbiome and associated metabolomic changes in patients with non-alcoholic fatty liver disease (NAFLD) and fibrosis who receive faecal microbiota transplant (FMT). The main questions is aims to answer is:

* To what extent is the gut microbiome transferable from donor to recipient in patients with NAFLD with fibrosis who receive FMT?
* What are the dynamics of how the gut microbiome changes over time in these patients?
* To what degree does the recipient metabolome change in association with this?

Participants will receive up to three capsulised FMT preparations prepared from a donor selected rationally based upon their metabolomic characteristics. They will be asked to attend for serial clinical assessments (including FibroScan and MRE/ MRI-PDFF), and will also be asked to provide serial blood, urine and stool samples for assessment of microbiome and metabolome profiling.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years of age.
2. Previously-diagnosed NAFLD, with predicted fibrosis based upon non-invasive assessment with FibroScan (i.e. liver stiffness measurement (LSM) > 8kPa).
3. Raised liver ALT (> 30IU/l for men, > 19IU/l for women) or AST (> 37IU/l for men, > 31IU/l for women) with negative non-invasive liver screen (including negative screen for viral hepatitis, autoimmune liver disease and metabolic liver disease, and normal echocardiogram within two years in the scenario where congestive hepatopathy may be considered).
4. Able to consent for themselves in English.

Exclusion Criteria:

1. Severe or life-threatening food allergy.
2. Pregnant or lactating women; or women trying to conceive.
3. Patients with suspected or confirmed cirrhosis (as assessed by clinical, radiological or histological criteria).
4. Use of particular medications, including:

   1. Systemic antibiotics within the six weeks prior to study enrolment.
   2. Immunosuppression that may influence risks related to FMT (including - but not limited to: use of corticosteroids within eight weeks of intervention; use of cytotoxic chemotherapy; use of azathioprine, tacrolimus, mycophenolate mofetil and/or immunosuppressive biologic therapy, e.g. infliximab).
   3. Use of GLP-1 agonists.
5. Patients not expected to survive the duration of the study's follow-up (six months).
6. Swallowing difficulties that may preclude safe use of FMT capsules, including oral-motor dyscoordination.
7. Alcohol consumption > 20g/ day.
8. Any active cancer (including treatment within the past six months).
9. Active infection at the point of recruitment, including COVID-19 infection.
10. Prior receipt of a liver transplant.
11. BMI < 23 in Asian potential participants and BMI < 25 in Caucasians.
12. Advanced chronic kidney disease (eGFR < 30 ml/min).
13. Chronic intestinal disease, including coeliac disease, cystic fibrosis, inflammatory bowel disease, irritable bowel syndrome, and chronic diarrhoea.
14. Prior bariatric surgery.
15. Patients unable to undergo MRI scans (e.g. due to the individual having metallic implants).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Change in faecal microbiome composition | 24 weeks after initial FMT
  Using 16S rRNA gene sequencing and shotgun metagenomic sequencing
Change in gut microbial metabolite composition | 24 weeks after initial FMT
  Using 1H-NMR and mass spectrometry

SECONDARY OUTCOMES:
Changes in liver fat on MRI | 16 weeks after initial FMT
  Using MRI-PDFF
Changes in liver fat on FibroScan | 16 weeks after initial FMT
  Using CAP
Changes in liver stiffness on MRI | 16 weeks after initial FMT
  Using MRE
Changes in liver stiffness on FibroScan | 16 weeks after initial FMT
  Using transient elastography
Changes in HbA1c | 24 weeks after initial FMT
Changes in insulin resistance | 24 weeks after initial FMT
  Combining fasting glucose and insulin levels to generate HOMA-IR
Changes in BMI | 24 weeks after initial FMT
  Through combination of measurement of weight in kilogram and height in metres, reporting BMI in kg/m^2
Changes in lipid metabolism | 24 weeks after initial FMT
  Serum lipid profile

CONTACTS AND LOCATIONS:
Overall Officials: Pinelopi Manousou, MD PhD, Principal Investigator — Imperial College London
Locations (1):
- Division of Digestive Diseases/ Liver Unit, St Mary's Hospital Campus, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only anonymised microbiome and metabolome data will be shared with other researchers via open access repositories

REFERENCES:
- [Derived] Aghara H, Patel M, Chadha P, Parwani K, Chaturvedi R, Mandal P. Unraveling the Gut-Liver-Brain Axis: Microbiome, Inflammation, and Emerging Therapeutic Approaches. Mediators Inflamm. 2025 Jun 18;2025:6733477. doi: 10.1155/mi/6733477. eCollection 2025. PMID 40568349